CLINICAL TRIAL: NCT06854913
Title: Impact of Orthopedic Surgery on Workers' Sleep
Acronym: ORTHOSLEEP
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Campus Bio-Medico (Other)
Responsible Party: Principal Investigator, Umile Giuseppe Longo, Professor, Fondazione Policlinico Universitario Campus Bio-Medico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 270.24 CET2 cbm; PNC0000007 - CUP: B53C22006980 (Other Grant/Funding Number: Italian Ministry of Research, under the complementary actions to the NRRP "Fit4MedRob - Fit for Medical Robotics")
Record Dates: First submitted 2025-02-12; First posted 2025-03-03 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Shoulder Musculoskeletal Disorders
Keywords: Musculoskeletal disorders; Shoulder pain; Sleep Monitoring; Orthopedic Surgery Outcomes; Wearable Sensors
MeSH Terms: conditions — Musculoskeletal Diseases; Shoulder Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Workers with shoulder musculoskeletal disorders (Experimental): Workers with shoulder musculoskeletal disorders will be enrolled from the Unit of Traumatology and Sports Medicine of FPUCBM. Patients who meet the inclusion criteria will be provided with an explanation of the study and the experimental protocol.
  After consenting to participate in the study and signing the informed consent, demographic and anthropometric data will be collected and registered on a database shared among authorized investigators involved in the project. In addition, patients will receive detailed verbal and written instructions on how to use the Medtronic Zephyr BioPatch™ wearable biosensor (Medtronic, Inc., Annapolis, MD, USA) for sleep monitoring. They will also be trained on how to complete the Consensus Sleep Diary, which they will fill out each morning after using the sensor.
  Sleep monitoring will be conducted at three key time points to assess changes in sleep patterns during the study. The first assessment will occur over two consecutive nights prior to surgery,
  Interventions: Other: Post-Operative monitoring using wearable biosensor; Other: Usability Assessment and Patient Willingness to Use Technology Description

INTERVENTIONS:
Other: Post-Operative monitoring using wearable biosensor — The protocol involves the use of the Medtronic Zephyr BioPatch™, a wearable biosensor, to monitor sleep quality and patterns in patients recovering from shoulder surgery. The device tracks physiological signals (ECG, HRV, respiratory rate) and postural changes, providing objective data on sleep profiles. Patients are assessed at three key time points: before surgery (baseline), two weeks after surgery (early recovery phase), and 30 days post-surgery (mid-recovery phase). The primary goal is to evaluate changes in sleep quality and patterns during the post-operative period, while also monitoring improvements in shoulder functionality and pain levels. This approach aims to provide insights into the relationship between sleep quality and recovery outcomes following shoulder surgery.
Other: Usability Assessment and Patient Willingness to Use Technology Description — The usability of the Medtronic Zephyr BioPatch™ is evaluated through patient feedback and questionnaires, focusing on comfort, ease of use, and reliability. Additionally, patient willingness to continue using the wearable sensor for sleep monitoring is assessed. This evaluation helps determine the practicality and acceptance of the technology in real-world rehabilitation settings, providing insights into its potential for long-term use in clinical practice.

SUMMARY:
Goal: The clinical investigation aims to evaluate the impact of orthopedic shoulder surgery on sleep quality and functional recovery in workers with shoulder musculoskeletal disorders. This will be assessed through validated questionnaires and physiological monitoring using wearable sensors.

Participant Population: The study will enroll at least 30 participants diagnosed with shoulder musculoskeletal disorders, such as rotator cuff tears, adhesive capsulitis, and glenohumeral osteoarthritis. Participants must be employed in physically demanding jobs that require frequent upper limb activity and are scheduled for orthopedic shoulder surgery.

Main Questions:

* How does post-operative rehabilitation influence sleep quality and functional recovery in workers with shoulder musculoskeletal disorders?
* To what extent does post-operative rehabilitation improve pain management and overall quality of life in these patients?
* How do patients perceive the usability and comfort of wearable sensors during their rehabilitation process?

Participant Tasks:

* Initial Assessment: Comprehensive clinical evaluation, including demographic and anthropometric data collection, and administration of the Pittsburgh Sleep Quality Index (PSQI).
* Wearable Sensor Training: Instruction on the proper use of the Medtronic Zephyr BioPatch™ wearable biosensor for monitoring physiological and postural signals.
* Sleep Monitoring: Participants will undergo sleep assessments at three key time points: Two nights before surgery (baseline measurement); Two weeks post-surgery during early rehabilitation; 30 days into the rehabilitation program.
* Daily Logging: Completion of the Consensus Sleep Diary each morning following sensor use.
* Functional Assessment: Objective evaluation of shoulder functionality through validated clinical scales and range of motion (ROM) assessments.
* Pain and Usability Evaluation: Measurement of pain reduction and usability of wearable technology using Patient-Reported Outcome Measures (PROMs).

DETAILED DESCRIPTION:
Shoulder pain represents one of the most widespread musculoskeletal issues globally, significantly impacting workers' quality of life and productivity. This condition often leads to substantial consequences for the overall health of affected individuals, with notable effects on essential aspects such as sleep. The majority of workers with shoulder pain also experience sleep disturbances, ranging from mild discomfort to complete inability to sleep. Nighttime pain, insomnia, and the inability to sleep on the affected side are factors that negatively impact patients' sleep quality. Poor sleep quality, in addition to pain, is one of the most common symptoms that drive patients to seek treatment and, if necessary, consider undergoing surgery.

Several studies have highlighted that rehabilitation following orthopedic surgery can significantly influence patients' sleep quality. Various patient-reported outcome measures (PROMs) have been introduced to assess improvements in sleep during the rehabilitation process. An example of a PROM is the Pittsburgh Sleep Quality Index (PSQI). With the growing interest in understanding the association between post-operative rehabilitation and sleep patterns, technologies have been introduced to provide objective and quantitative measures of these changes.

The gold standard for studying sleep is polysomnography, which, due to its intrusive nature, can alter the sleep quality and profile for reasons unrelated to the surgical rehabilitation itself. Recent studies have shown that wearable sensors measuring physiological parameters (e.g., ECG, HRV) and posture, combined with advanced artificial intelligence techniques, offer the possibility to monitor sleep profiles with good reliability in a non-intrusive and real-time manner.

This study aims to use non-invasive wearable sensors and artificial intelligence algorithms to monitor patients undergoing post-operative rehabilitation following shoulder surgery. The objective is to explore in-depth the variations in sleep patterns and quality during the rehabilitation process, analyzing the relationship between sleep and recovery. This research seeks to empirically demonstrate the benefits of post-operative rehabilitation on improving the sleep quality and profile of patients with shoulder disorders.

This research is of critical importance as it provides essential insights for clinicians and workers regarding the impact of rehabilitation on sleep quality. Understanding the relationship between shoulder pain, rehabilitation, and sleep disturbances is a key clinical issue. The outcomes of this study could have significant implications for the overall management of shoulder pain, potentially enhancing clinical practices and improving healthcare for individuals affected by these conditions. In addition, this research aims to offer valuable information that will inform optimal treatment strategies, ultimately enhancing workplace productivity and overall health.

ELIGIBILITY:
Inclusion Criteria

* Informed consent obtained.
* Age ≥ 18 years.
* Good understanding of spoken and written Italian.
* Diagnosis of shoulder musculoskeletal disorders.
* Employment in a physically demanding job requiring frequent upper limb activity.
* Workers scheduled to undergo orthopedic shoulder surgery.
* Workers who have accepted the surgical treatment.

Exclusion Criteria

* Patients with sleep disorders.
* Patients undergoing pharmacological treatments that could potentially affect sleep patterns (e.g., antidepressants, hypnotics, and stimulants).
* Failure to sign informed consent.
* Patients with neuromuscular diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Heart Rate Evaluation During Sleep Across Different Rehabilitation Phases | three key time points: before surgery (baseline), two weeks after surgery (early recovery phase), and 30 days post-surgery (mid-recovery phase)
  Heart rate will be monitored using wearable sensors during sleep across different rehabilitation phases. It will be recorded in beats per minute to evaluate the physiological response to recovery and adaptation throughout the rehabilitation process.
Respiratory Rate Evaluation Evaluation During Sleep Across Different Rehabilitation Phases | three key time points: before surgery (baseline), two weeks after surgery (early recovery phase), and 30 days post-surgery (mid-recovery phase)
  Respiratory rate will be monitored using wearable sensors during sleep across different rehabilitation phases. It will be recorded in breaths per minute to assess the physiological response to recovery and adaptation throughout the rehabilitation process
Change in Sleep Efficiency Across Different Rehabilitation Phases | three key time points: before surgery (baseline), two weeks after surgery (early recovery phase), and 30 days post-surgery (mid-recovery phase)
  Sleep efficiency is defined as the percentage of total sleep time (TST) relative to the total time spent in bed (sleep opportunity). It is calculated by dividing the amount of time spent asleep by the total time in bed and multiplying by 100. This measurement will be obtained using wearable sensors. Values of 85% or higher are generally considered indicative of good sleep quality. This parameter is critical for assessing how effectively the available time for sleep is used and for identifying sleep fragmentation or disruptions.
Change in Sleep Duration Across Different Rehabilitation Phases | three key time points: before surgery (baseline), two weeks after surgery (early recovery phase), and 30 days post-surgery (mid-recovery phase)
  Sleep duration refers to the total amount of time a subject spends asleep during the night, expressed in minutes or hours. It is measured from the onset of sleep until the final awakening, excluding periods of wakefulness. The wearable device continuously tracks sleep and wake states, providing an accurate account of total sleep time. For adults, a duration of 7 to 9 hours is typically recommended. Monitoring sleep duration is essential to evaluate the restorative quality of sleep and to compare changes across different rehabilitation phases.
Change in Wake After Sleep Onset (WASO) Across Different Rehabilitation Phases | three key time points: before surgery (baseline), two weeks after surgery (early recovery phase), and 30 days post-surgery (mid-recovery phase)
  WASO is defined as the total time, in minutes, that a subject remains awake after the initial onset of sleep and before the final awakening. A wearable device records all episodes of wakefulness during the sleep period and sums them to calculate WASO. A WASO value of less than 30 minutes is generally considered normal for healthy sleep. Elevated WASO values can indicate increased sleep fragmentation, which may compromise the quality of sleep.
Change in Sleep Latency Across Different Rehabilitation Phases | three key time points: before surgery (baseline), two weeks after surgery (early recovery phase), and 30 days post-surgery (mid-recovery phase)
  Sleep latency is the duration, measured in minutes, between the moment a subject goes to bed (or turns off the lights) and the onset of sleep. The wearable device identifies the sleep onset as the first epoch classified as sleep. A sleep latency of less than 20 minutes is generally considered normal, whereas prolonged sleep latency may signal difficulties in initiating sleep, possibly due to pre-surgical anxiety or post-surgical discomfort.

SECONDARY OUTCOMES:
Change in Sleep Data among different rehabilitation phases | Three key time points: before surgery (baseline), two weeks after surgery (early recovery phase), and 30 days post-surgery (mid-recovery phase).
  This outcome involves the use of the Consensus Sleep Diary, which patients complete each morning after using the Medtronic Zephyr BioPatch™. The diary collects information on sleep patterns, including bedtime, wake time, and perceived sleep quality.
Evaluation of the usability and Comfort of Wearable Technology | Three key time points: before surgery (baseline), two weeks after surgery (early recovery phase), and 30 days post-surgery (mid-recovery phase).
  This outcome evaluates the usability and comfort of the Medtronic Zephyr BioPatch™ using validated scales, such as the System Usability Scale (SUS). SUS is a standardized tool for assessing the ease of use and overall usability of the device. The total score ranges from 0 to 100, with 0 indicating poor usability and 100 indicating excellent usability. Higher scores represent a better outcome in terms of perceived usability of the system.
Evaluation of the Objective Improvement in Shoulder Functionality | Three key time points: before surgery (baseline), two weeks after surgery (early recovery phase), and 30 days post-surgery (mid-recovery phase).
  This outcome measures the improvement in shoulder functionality using range of motion (ROM) assessments. Shoulder ROM will be evaluated using stereophotogrammetric systems during the execution of movements of clinical relevance.
Evaluation of the Reduction in Pain Levels among different rehabilitation phases | Three key time points: before surgery (baseline), two weeks after surgery (early recovery phase), and 30 days post-surgery (mid-recovery phase).
  This outcome evaluates the reduction in pain using standardized pain assessment tools, such asthe Visual Analog Scale (VAS). VAS is a self-reported measure of pain intensity, ranging from 0 (no pain) to 10 (worst pain imaginable).

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Campus Bio-Medico, Rome, Italy, Italy

IPD SHARING:
Plan to Share IPD: Yes
The ownership of the data is of the promoter and shared with the investigators and will be managed according to the agreements between the participating institutions and with the researchers. Data Property belongs to Fondazione Policlinico Universitario Campus Bio-Medico. The personnel involved in this study will have access to all data. In agreement with the ICH-GCP, the principal investigator of the study agrees to produce a report on the study, share all the data collected as described in the Protocol, and ensure that the data are reported responsibly and consistently.
  The transmission or dissemination of data through scientific publications and/or presentations in congresses, conferences, seminars, and participation in multicenter studies will take place exclusively following a purely statistical processing of the same, or in any case, in an anonymous form.